CLINICAL TRIAL: NCT00844129
Title: Spinal Abnormalities in Neurofibromatosis Type 1 (NF1)
Acronym: Spine
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, David Viskochil, Professor, University of Utah
Other Study IDs: 15464; R01NS050509 (NIH)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Neurofibromatosis Type 1
Keywords: neurofibromatosis type 1; spinal abnormalities; scoliosis
MeSH Terms: conditions — Neurofibromatosis 1; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurofibromatosis Type 1: Children with Neurofibromatosis Type 1

SUMMARY:
The purpose of this study is to determine the incidence and clinical history of neurofibromatosis type 1-related spinal abnormalities.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is a common genetic disorder that is associated with spinal abnormalities which are varied and may include scoliosis, neurofibromas, meningoceles, and vertebral defects. Skeletal abnormalities occur in more than one third of individuals with the disorder. These abnormalities are unpredictable and the pathogenesis, natural history, and clinical outcome remain relatively unclear.

The primary objective of this study is to determine the incidence and clinical history of NF1-related spinal abnormalities in children with NF1, over a 3-year period.

In the study, researchers will enroll children between ages 6 and 9 years who have been diagnosed with NF1 to look at changes in the spine. Participants in the study will be followed yearly for a total of 4 evaluations. Evaluations may include bone scans, spinal x-rays, magnetic resonance imaging (MRI), computed tomography (CT) scans, and urine samples.

Information gained from this study may lead to a better understanding of the causes of bone disease in NF1, and improved treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NF1
* Age greater than 6 years at time of enrollment
* Age less than 9 year and 1 day at time of enrollment
* Tanner Stage not greater than 1

Exclusion Criteria:

* Prior surgical repair of spine
* Short-segment (4-6 vertebrae) curve with a Cobb angle of 45°or more
* Hormone replacement therapy
* Chronic steroid use
* Tibial pseudarthrosis
* Other chronic medical problems known to influence bone health (i.e. diabetes mellitus, cerebral palsy, etc.)

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The cohort will be recruited from a primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Scoliosis and it's progression | 4 years

SECONDARY OUTCOMES:
Differences in other bone health variables as measured by thoracic MRIs, Dexa (xray measuring bone density), pQCT (a cross sectional picture of the tibia), urine analysis, and scoli series (xrays to look for scoliosis). | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: David Viskochil, MD, PhD, Principal Investigator — Division of Medical Genetics, Department of Pediatrics, University of Utah
Locations (1):
- University Health Care, 50 North Medical Drive, Salt Lake City, Utah, United States